CLINICAL TRIAL: NCT03817216
Title: Prostatic Urethral Lift (PUL) Pre-/Post-Radiation Treatment for Prostate Cancer: Prospective Analysis of Outcomes in Patients With Obstructive Urinary Symptoms
Brief Title: Prostatic Urethral Lift (PUL) Pre-/Post-Radiation Treatment for Prostate Cancer
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: re-written and submitted as a new study
Sponsor: Case Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: CASE10818
Record Dates: First submitted 2018-12-04; First posted 2019-01-25 (Actual); Last update posted 2020-03-12 (Actual); Status verified 2020-03

CONDITIONS: Benign Prostatic Hyperplasia (BPH); Prostate Cancer
Keywords: Prostatic Urethral Lift (PUL)
MeSH Terms: conditions — Prostatic Hyperplasia; Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (3):
- Prostatic Urethral Lift (PUL) post-EBRT (Experimental): Prostatic Urethral Lift (PUL) following External Beam Radiotherapy (EBRT)
  Interventions: Device: Prostatic Urethral Lift (PUL)
- Prostatic Urethral Lift (PUL) pre-BT (Experimental): Prostatic Urethral Lift (PUL) preceding Brachytherapy (BT)
  Interventions: Device: Prostatic Urethral Lift (PUL)
- Prostatic Urethral Lift (PUL) post-BT (Active Comparator): Prostatic Urethral Lift (PUL) following Brachytherapy (BT)
  Interventions: Device: Prostatic Urethral Lift (PUL)

INTERVENTIONS:
Device: Prostatic Urethral Lift (PUL) — PUL/ UroLift® is an FDA-approved device for the treatment of obstructive symptoms due to benign prostatic hyperplasia (BPH). This study evaluates UroLift's efficacy participants with obstructive symptoms who are candidates for radiotherapy or those who developed obstructive symptoms after radiotherapy.

SUMMARY:
The purpose of this study is to test the use of the Prostatic Urethral Lift (PUL), Urolift®, in prostate cancer (Pca) participants seeking or undergoing radiotherapy for relief of urinary obstructive symptoms.

DETAILED DESCRIPTION:
Prostatic Urethral Lift (PUL)/ UroLift® is an FDA-approved device for the treatment of obstructive symptoms due to benign prostatic hyperplasia (BPH) (also called prostate gland enlargement). This study seeks to evaluate UroLift's efficacy in a unique cohort of participants with obstructive symptoms who are candidates for radiotherapy or those who developed obstructive symptoms after radiotherapy. The primary objective of this study is to achieve urinary obstructive symptom relief in prostate cancer participants undergoing radiotherapy treatment with placement of PUL. This will be quantified using primary effectiveness endpoints:

* For PUL placement post-EBRT and post-BT: ≥ 30% or ≥ 4 point International Prostate Symptom Score (IPSS) reduction 3 months after PUL.
* For PUL placement pre-BT: ≥ 30% or ≥ 4 point IPSS reduction 3 months after Brachytherapy (BT) from pre-PUL baseline.

The team will also assess participant outcomes with regard to International Prostate Symptom Score (IPSS), peak urine flow (Qmax),post-void residual (PVR), quality of life (QOL) scores, Benign Prostatic Hyperplasia Impact Index (BPHII) scores, Men's Sexual Health Questionnaire (MSHQ) scores, and urinary incontinence at 6 and 12 months of PUL placement post-External Beam Radiotherapy (EBRT), post-BT, and pre-BT.

ELIGIBILITY:
Inclusion Criteria:

* International Prostate Symptom Score ≥ 12.
* Peak flow rate ≤ 12 ml/sec with at least 125 ml voided urine.
* Prostate volume ≤ 80 cc as measured either by trans-rectal ultrasound (US) or Magnetic Resonance Imaging (MRI).

Exclusion Criteria:

* Obstructive median lobe of the prostate.
* Active urinary tract infection.
* Neurogenic non-obstructive voiding dysfunction.
* Obstructive symptoms secondary to prostate cancer (via cystoscopy).
* Patients with prior Transurethral resection of the prostate (TURP).
* Patients with prior history of urethral stricture.

Min Age: 51 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-12 (Estimated); Primary Completion 2022-06-30 (Estimated); Study Completion 2023-03-30 (Estimated)

PRIMARY OUTCOMES:
Mean change in International Prostate Symptom Score (IPSS) - Arms: PUL placement post-EBRT and PUL placement post-BT | 3 months post-PUL placement
  IPSS is an eight-question written screening tool used to screen for, rapidly diagnose, track the symptoms of, and suggest management of the symptoms of benign prostatic hyperplasia.
  A mean change in International Prostate Symptom Score (IPSS) will be considered effective if the following condition is met:
  ≥ 30% or ≥ 4 point IPSS reduction 3 months after PUL.
Mean change in International Prostate Symptom Score (IPSS) - Arm: PUL placement pre-BT. | 3 months post-BT
  IPSS is an eight-question written screening tool used to screen for, rapidly diagnose, track the symptoms of, and suggest management of the symptoms of benign prostatic hyperplasia.
  A mean change in International Prostate Symptom Score (IPSS) will be considered effective if the following condition is met:
  * 30% or ≥ 4 point IPSS reduction 3 months after BT from pre-PUL baseline.

SECONDARY OUTCOMES:
Mean change in International Prostate Symptom Score (IPSS) | 6 and 12 months post-BT (pre-BT arm) or post-PUL placement (Post-BT & Post-EBRT arms)
  IPSS is an eight-question written screening tool used to screen for, rapidly diagnose, track the symptoms of, and suggest management of the symptoms of benign prostatic hyperplasia.
  Mean change in IPSS score will be reported
Mean change in peak urinary flow rate (Qmax) | 6 and 12 months post-BT (pre-BT arm) or post-PUL placement (Post-BT & Post-EBRT arms)
  Qmax is the quantity of urine measured over a specified period of time. A significant outcome would be a greater than 50% change in Qmax.
Quality of life scores from last question on IPSS questionnaire | 6 and 12 months post-BT (pre-BT arm) or post-PUL placement (Post-BT & Post-EBRT arms)
  QOL score (last question in the IPSS questionnaire): If you were to spend the rest of your life with your urinary condition just the way it is now, how would you feel about that?
  With answer options on a 0-6 scale with 0 being delighted and 6 being terrible.
Mean change in Benign Prostatic Hyperplasia Impact Index (BPHII) scores | 6 and 12 months post-BT (pre-BT arm) or post-PUL placement (Post-BT & Post-EBRT arms)
  The Benign Prostatic Hyperplasia Impact Index (BPHII) is a self-administered questionnaire with four questions about urinary problems during the past month regarding physical discomfort, worry about health, how bothersome symptoms are, and whether the symptoms are interfering with doing usual activities.
  Mean change in BPHII score will be reported.
Mean change in the MSHQ total score | 6 and 12 months post-BT (pre-BT arm) or post-PUL placement (Post-BT & Post-EBRT arms)
  Men's Sexual Health Questionnaire (MSHQ) is a 18-item questionnaire focused on assessing three core function domains (erection, ejaculation and satisfaction).
  Mean change in the MSHQ ejaculation total score will be reported.
Urinary incontinence measured by number of pads used | 6 and 12 months post-BT (pre-BT arm) or post-PUL placement (Post-BT & Post-EBRT arms)
  Assessment of urinary incontinence associated with the procedure measured by change number of pads used per day.
Urinary incontinence measured by quality of stress or urge | 6 and 12 months post-BT (pre-BT arm) or post-PUL placement (Post-BT & Post-EBRT arms)
  Assessment of urinary incontinence associated with the procedure as measured by quality: stress or urge.
Urinary incontinence measured by cough stress test | 6 and 12 months post-BT (pre-BT arm) or post-PUL placement (Post-BT & Post-EBRT arms)
  Assessment of urinary incontinence associated with the procedure as measured by cough test.
Urinary incontinence measured by time to resolve | 6 and 12 months post-BT (pre-BT arm) or post-PUL placement (Post-BT & Post-EBRT arms)
  Assessment of urinary incontinence associated with the procedure as measured by time to resolve.
Mean change in post-void residual (PVR) | 3, 6, and 12 months post-BT (pre-BT arm) or post-PUL placement (Post-BT & Post-EBRT arms
  Assessment of PVR, the amount of urine left in the bladder after urination.

CONTACTS AND LOCATIONS:
Overall Officials: Irina Jaeger, MD, Principal Investigator — University Hospitals Cleveland Medical Center